CLINICAL TRIAL: NCT04740099
Title: Surviving Opioid Overdose With Naloxone Education and Resuscitation Trial (SOONER): Randomized Trial and Embedded Qualitative Study to Compare the Effectiveness of point-of Care Overdose Education and Naloxone Distribution Versus Referral to an Existing Community Program in the Management of Simulated Opioid-associated Resuscitative Emergencies.
Brief Title: Surviving Opioid Overdose With Naloxone Education and Resuscitation Trial (SOONER)
Acronym: SOONER
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study never started due to COVID-19.
Sponsor: Unity Health Toronto (Other)
Collaborators: Toronto Public Health (Other Government); Ontario College of Art and Design (OCAD) (Unknown); University of Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 19-169
Record Dates: First submitted 2019-09-04; First posted 2021-02-05 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Opioid Use; Opioid-Related Disorders; Opioid Withdrawal; Opioid Overdose; Education; Resusitation
MeSH Terms: conditions — Opioid-Related Disorders; Opiate Overdose | interventions — Receptor Protein-Tyrosine Kinases; Standard of Care

STUDY DESIGN:
Intervention Model Description: Pragmatic, multi-site, 2-armed, parallel-group, best available care controlled, analyst- and outcome assessor-blinded, superiority trial with embedded qualitative study.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SOONER Training (Intervention) (Experimental): Arm receives video training and kit designed by SOONER team.
  Interventions: Other: SOONER Video & Kit
- Standard of care training (control) (Other): Participant referred to standard of care (community based Naloxone training)
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: SOONER Video & Kit — A brief animated video including basic instructions for opioid overdose response accompanied by a Naloxone kit with an info graphic.
  Other Names: SOONER Naloxone kit
  Arms: SOONER Training (Intervention)
Other: Standard of Care — A handout including a map and list of locations offering this service.
  Other Names: Community Based Naloxone training referral
  Arms: Standard of care training (control)

SUMMARY:
Among people at risk of opioid overdose and receiving care in an academic emergency department, family practice, opioid substitution clinic or general inpatient units, does brief opioid overdose resuscitation training and naloxone distribution reduce resuscitation failures in a simulated overdose even, in comparison with standard-of-care referral to a local OEND program, within 14 days post-intervention? Can an integrated participant recruitment and retention strategy recruit approximately 28 eligible participants within 4 weeks and maintain less than 50% attrition rates in the context of a randomized trial on point-of-care OEND and simulated overdose resuscitation performance in family practice, emergency department, and addictions settings?

ELIGIBILITY:
Inclusion Criteria:

1. adults ≥16 years of age, and
2. Eligible for overdose education according to criteria adapted from the 2015 American Heart Association Guidelines by meeting any one or more of the following criteria:

   1. has a history of taking opioids at recognized 'high doses' (whether by prescription or otherwise, defined as >100mg morphine equivalent per day);
   2. has required emergency care for opioid overdose previously;
   3. is enrolled in opioid agonist treatment programs, including methadone or buprenorphine maintenance programs, or stopped an opioid agonist treatment program in the last 6 months;
   4. uses non-medical opioids, injects opioids, or acquires opioids from sources other than a pharmacy or healthcare setting;
   5. has a history of non-medical opioid use who are being released from prison;
   6. is receiving prescription opioid therapy with risk factors for adverse effects, including i. relevant comorbidities, ii. co-prescriptions of benzodiazepines or other sedatives, iii. concomitant ongoing alcohol use, iv. use of prescription opioids not as prescribed.
   7. is likely to witness an opioid overdose, defined as anyone who lives with or is in frequent contact with others who use opioids, or who has previously witnessed an opioid overdose.

Exclusion Criteria:

1. plan to move away from Toronto during the study period
2. have no mode of contact or follow-up,
3. have a community do not resuscitate order,
4. have a terminal illness, end-of-life care, or illness likely to result in death within the study period,
5. are an active or previously practicing healthcare professional or professional first responder (e.g.: firefighter, police officer, lifeguard, industrial first responder), or
6. have insufficient English language skills to participate in the study.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Satisfactory basic life support performance | 4-14 days after enrolment
  Satisfactory basic life support performance on a standardized high fidelity overdose simulation, as assessed by the consensus of two trained clinicians.

SECONDARY OUTCOMES:
Performance on basic resuscitation skill: Recognize the Emergency | 4-14 days after enrolment
  Skill performance will be rated as either satisfactory or unsatisfactory by two trained clinicians. Inter-rater reliability of the assessors for each of the eight secondary outcome skills will be calculated.
Performance on basic resuscitation skill: Position the Victim | 4-14 days after enrolment
  Skill performance will be rated as either satisfactory or unsatisfactory by two trained clinicians. Inter-rater reliability of the assessors for each of the eight secondary outcome skills will be calculated.
Performance on basic resuscitation skill: Activate emergency medical services | 4-14 days after enrolment
  Skill performance will be rated as either satisfactory or unsatisfactory by two trained clinicians. Inter-rater reliability of the assessors for each of the eight secondary outcome skills will be calculated.
Performance on basic resuscitation skill: Administer Naloxone | 4-14 days after enrolment
  Skill performance on device preparation and correct administration will be rated as either satisfactory or unsatisfactory by two trained clinicians. Inter-rater reliability of the assessors for each of the eight secondary outcome skills will be calculated.
Performance on basic resuscitation skill: Hand placement | 4-14 days after enrolment
  Skill performance will be rated as either satisfactory or unsatisfactory by two trained clinicians. Inter-rater reliability of the assessors for each of the eight secondary outcome skills will be calculated.
Performance on basic resuscitation skill: chest compressions | 4-14 days after enrolment
  Skill performance (rate and depth of chest compressions) will be rated as either satisfactory or unsatisfactory by two trained clinicians. Inter-rater reliability of the assessors for each of the eight secondary outcome skills will be calculated.
Performance on basic resuscitation skill: continue compressions until end of simulation | 4-14 days after enrolment
  Skill performance will be rated as either satisfactory or unsatisfactory by two trained clinicians. Inter-rater reliability of the assessors for each of the eight secondary outcome skills will be calculated.
Performance on basic resuscitation skill: order of operations | 4-14 days after enrolment
  Skill performance will be rated as either satisfactory or unsatisfactory by two trained clinicians. Inter-rater reliability of the assessors for each of the eight secondary outcome skills will be calculated.

OTHER OUTCOMES:
Standardized assessor-implemented survey and interview responses to measure overdose-related knowledge and behaviours | 4-14 days after enrolment
  The questionnaires were developed for the Toronto Public Health OEND program evaluation using data points from other overdose education and naloxone distribution programs and from the validated Opioid Overdose Knowledge and Attitudes Scales (OOKS and OOAS). We also included relevant questions from a national survey of injection drug users (ITRACK, Health Canada) and the CAMH Monitor conducted by the Centre for Addiction and Mental Health (CAMH). The questionnaire items include:
  1. Demographics: age, gender, ethnicity, housing status, and neighbourhood
  2. Prescription medications
  3. Opioid and non-opioid drug use in past 4 weeks: drug, amount, route, frequency
  4. Drug use setting: where and with whom opioids were used
  5. Periods of abstinence
  6. Use of prevention strategies, and speaking to others about overdose or overdose response
  7. Knowledge of overdose and naloxone use
  8. Status of naloxone kit
  9. Willingness and confidence to respond to overdose

CONTACTS AND LOCATIONS:
Overall Officials: Carol Strike, PhD, Principal Investigator — University of Toronto; Aaron Orkin, MD, Study Chair — University of Toronto
Locations (1):
- St. Michael's Hospital, Unity Health Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
All publications will indicate that original de-identified study data and statistical coding is available upon request from the Steering Committee. This information and will be shared freely with corresponding scholars and the public, on request.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Available on an ongoing basis upon request
Access Criteria: At the discretion of the research team